CLINICAL TRIAL: NCT03793491
Title: Study About Personality, as a Predictive Factor of Therapeutic Response on Quality of Life After Continuous Perfusion of Dopaminergic Drugs (by Subcutaneous Apomorphine Infusion or Intrajejunal Infusion of Levodopa-carbidopa), in Parkinson's Disease
Brief Title: Personality, as a Predictive Factor of Therapeutic Response on Quality of Life After Continuous Perfusion of Dopaminergic Drugs, in Parkinson's Disease
Acronym: PSYCHO-PERF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/18/0390
Record Dates: First submitted 2018-12-21; First posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Parkinson Disease
Keywords: continuous infusion; personality
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having Parkinson's disease: Parkinson's patients presenting motor fluctuations and/or disabling dyskinesia and in need of the establishment of a second line treatment by subcutaneous apomorphine infusion or intrajejunal infusion of levodopa-carbidopa in the context of classical care of their Parkinson's disease. Patients will have TCI scale and PDQ-39 scale.
  Interventions: Other: TCI scale; Other: PDQ-39 scale

INTERVENTIONS:
Other: TCI scale — TCI scale : Evaluation of the patient's personality with the TCI before that the treatment by continuous infusion started.
  Other Names: Temperament and Character Inventory scale (TCI); Quality of life scale
Other: PDQ-39 scale — PDQ-39 scale: Comparison of life quality before and after the starting of he treatment by continuous infusion.
  Other Names: Parkinson's Disease Questionnaire (PDQ-39)

SUMMARY:
The aim of the study is to evaluate if patients' personality could be considerate as predictive factor of quality of life after the establishment of continuous infusion of dopaminergic treatments to observe if there are predictive personality's profiles of specific therapeutic response (Deep Brain Stimulation (DBS) of the subthalamic nucleus (STN) or continuous infusion).

DETAILED DESCRIPTION:
Parkinson's disease leads to quality of life degradation, especially at level of motor complications. Second line treatment can be proposed to patients. There are deep brain stimulation and two treatments by continuous perfusion: subcutaneous apomorphine infusion and intrajejunal infusion of levodopa-carbidopa. These treatments allow improvement of end-of-dose akinesia, dyskinesia, and a diminution of treatments per os. Nonetheless, they also lead to some side effects and complications. Currently, there are no scientific data to compare the efficacy of these two techniques on motor and non-motor symptoms. Choice is made according to the profile of the patient mainly based on side effects risks, and practitioner's habits. There are still no predictive factors clearly defined to judge of the best efficacy of these treatments according to the patients. Moreover, in an additional study named PSYCHO-STIM, the investigator have discovered that personality can be a predictive factor of quality of life amelioration 1 year after deep brain stimulation. It's why the investigator would like to test personality as a predictive factor of therapeutic response after both continuous perfusions that are available for the patients. Thus, patients beginning a treatment by subcutaneous apomorphine infusion or intrajejunal infusion of levodopa-carbidopa will be included. The investigator will evaluate their personality with the questionnaire "TCI" (Temperament and Character Inventory) and the investigator will assess their quality of life (PDQ-39), looking for the percentage of amelioration 6 months after the treatment by continuous infusion started. As secondary criteria, depression (HAMD), anxiety (HAMA), apathy (LARS), motility (MDS-UPDRS) and clinic severity (CGIS) will also be accessed before the treatment change and six months later.

ELIGIBILITY:
Inclusion Criteria:

* Patients having Parkinson's disease according to United Kingdom Parkinson's Disease Society Brain Bank (UKPDSBB) criteria
* All Parkinson's patients presenting motor fluctuations and/or disabling dyskinesia and in need of the establishment of a second line treatment by subcutaneous apomorphine infusion or intrajejunal infusion of levodopa-carbidopa in the context of classical care of their Parkinson's disease
* Patient able to give its free and informed consent
* Patient having a social security

Exclusion Criteria:

* Patients presenting atypical Parkinson's syndrome
* Patients having a deep brain stimulation
* Patient having a psychiatric disease such as: mood disorders, psychotic disorder…
* Patients presenting a cognitive decline evaluated by a Montreal Cognitive Assessment (MoCA) score inferior to 24
* None ability to give its consent
* Patients unable to realize the tests provided in the context of this study
* Patients under supervision, curators, or legal guardian
* Patients non-affiliated to a social security
* Patients in exclusion period of another study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-12-18 (Estimated); Study Completion 2021-06-18 (Estimated)

PRIMARY OUTCOMES:
percent of improvement of quality of life score at 6 months after the beginning of the second line treatment | day 1
  Evaluation of life quality using Parkinson's Disease Questionnaire (PDQ-39) scale before (day 1) and after (6 month) the starting of perfusion treatment
percent of improvement of quality of life score at 6 months after the beginning of the second line treatment | 6 months
  Evaluation of life quality using PDQ-39 scale before and after the starting of perfusion treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chrisitine BREFEL COURBON, PH, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No